CLINICAL TRIAL: NCT06410729
Title: Significance of Benign Lymph Node Enlargement in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2020123
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Benign mesenteric lymph node enlargement (BLNE): Lymph nodes with a diameter > 8 mm on preoperative imaging without metastasis on postoperative pathology were termed benign mesenteric lymph node enlargement.
  Interventions: Other: Observational study, no intervention
- Non-benign mesenteric lymph node enlargement (NBLNE): Lymph nodes with a diameter < 8 mm on preoperative imaging without metastasis on postoperative pathology were termed non-benign mesenteric lymph node enlargement.
  Interventions: Other: Observational study, no intervention
- Metastatic mesenteric lymph node enlargement (MLNE): Lymph nodes with a diameter > 8 mm on preoperative imaging with metastasis on postoperative pathology were termed metastatic mesenteric lymph node enlargement .
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention

SUMMARY:
The objective of this observational study was to investigate the clinical significance of benign mesenteric lymph node （BLNE） enlargement in patients with colorectal cancer. The main questions it aims to answer are:

Do patients with benign mesenteric lymph node enlargement have a better prognosis? What are the clinical characteristics of benign mesenteric lymph node enlargement? As part of routine medical care for colorectal cancer, we will follow up with all participants over the course of the study.

DETAILED DESCRIPTION:
From January 2015 to June 2023, 2,270 patients with colorectal cancer received surgical treatment at Peking University Third Hospital. The clinical data of these patients were recorded retrospectively and the eligible patients were divided into two groups. According to the 9th edition of the TNM staging System published by the AJCC, the BLNE group included the mesenteric BLNE group, while the non-benign lymph node enlargement (NBLNE) group was the control group. Inclusion criteria were :1) No regional lymph node metastasis or distant metastasis; 2) Stage I and II patients with AJCC staging system; 3) Radical CRC resection reached R0 status, no positive lymph nodes; Colonoscopy confirmed a single malignant lesion. Exclusion criteria :1) emergency surgery or preoperative complications such as intestinal obstruction and perforation; 2) Positron emission tomography (PET-CT) suspected distant metastasis; 3) Preoperative neoadjuvant therapy; 4) Hereditary colorectal cancer such as familial adenomatous polyposis; Microsatellite instability (MSI) was confirmed by pathology. In early colorectal cancer, MSI-H status is associated with a favorable prognosis and enhanced anti-tumor immune response. Therefore, we excluded these patients to avoid their influence on prognosis. 6) Lack of imaging data; 7) Loss of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* no regional lymph node metastasis or distant metastasis;
* stage I and II patients in the AJCC staging system;
* radical CRC resection achieving R0 status with no positive lymph nodes;
* a single malignant lesion confirmed via colonoscopy

Exclusion Criteria:

* underwent emergency surgery or had preoperative complications such as intestinal obstruction or perforation;
* had suspected distant metastasis on positron emission tomography (PET-CT);
* received preoperative neoadjuvant therapy;
* had hereditary CRC such as familial adenomatous polyposis;
* had microsatellite instability (MSI) confirmed by pathology.
* lacked imaging data;
* were lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone radical colorectal cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 2270 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival of participants | The time from the participants' first postoperative day to their last follow-up.
  From the time participants started undergoing radical surgery until their tumors returned or they died from tumor causes. The unit is month.

SECONDARY OUTCOMES:
Overall survival of the participants | The time from the participants' first postoperative day to their last follow-up.
  The time from the time participants began undergoing radical surgery until they died from any cause. Unit is month.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Wang, M.D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided